CLINICAL TRIAL: NCT03780634
Title: Hepatic Artery Infusion Chemotherapy Plus Programmed Cell Death Protein-1 (PD-1) Antibody vs Hepatic Artery Infusion Chemotherapy Plus Sorafenib for Advanced Hepatocellular Carcinoma
Brief Title: HAIC Plus PD-1 Antibody vs HAIC Plus Sorafenib for Advanced HCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S059
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatic arterial infusion chemotherapy; Programmed cell death protein-1 antibody; Oxaliplatin, 5-Fluorouracil and Leucovorin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — spartalizumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC plus PD-1 antibody (Experimental): Participants received PD-1 antibody intravenously and hepatic artery infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin every 3 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Procedure: HAIC; Drug: PD-1 antibody
- HAIC plus sorafenib (Active Comparator): Participants received sorafenib capsules 400mg bid in continuous 21-day treatment cycles, and received hepatic artery infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin every 3 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Procedure: HAIC; Drug: Sorafenib

INTERVENTIONS:
Procedure: HAIC — administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 3 weeks
Drug: PD-1 antibody — 200mg intravenously every 3 weeks
  Other Names: Programmed cell death 1 antibody
  Arms: HAIC plus PD-1 antibody
Drug: Sorafenib — 400 mg Bid Po
  Arms: HAIC plus sorafenib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic artery infusion chemotherapy (HAIC) combined with Programmed Cell Death Protein-1 (PD-1) antibody compared with HAIC plus sorafenib in patients with advanced hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
The results of our preliminary pilot study suggested that sorafenib combined with hepatic arterial infusion chemotherapy (HAIC) may improve the survivals for advanced hepatocellular (HCC). Programmed Cell Death Protein-1 (PD-1) antibody has been proved effective and safety for advanced HCC. There is no study about HAIC plus PD-1 antibody. Thus, the investigators carried out this prospective randomized control study to compare HAIC plus sorafenib and HAIC plus PD-1 antibody.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Major portal vein tumor thrombus (Vp3,Vp4)
* Eastern Cooperative Oncology Group performance status of 0 to 1
* with no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection, local ablative therapy and any other cured treatment.
* The following laboratory parameters:

  * Platelet count ≥ 75,000/μL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 30mmol/L
  * Serum albumin ≥ 30 g/L
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or PT/APTT within normal limits
  * Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1), or date of death, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on RECIST.
Adverse Events | 12 months
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospital, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong